CLINICAL TRIAL: NCT01373463
Title: A Phase I Trial of Preoperative Carboplatin or Cisplatin and Pemetrexed With Thoracic Radiation Therapy Followed by Lobectomy in Resectable Stage III Patients With Non-Squamous Non Small Cell Lung Cancer (NSCLC)
Brief Title: Cisplatin and Pemetrexed With Radiation Followed by Lobectomy
Acronym: CisPemXetSrg
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left site
Sponsor: Medical University of South Carolina (Other)
Responsible Party: George Simon, MD, Hollings Cancer Cetner Medical University of South Carolina
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 101466
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Nonsquamous Nonsmall Cell Neoplasm of Lung; Nonsmall Cell Lung Cancer Stage III
Keywords: resectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Radiotherapy; Cisplatin; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): 1. Patients will be given the drugs pemetrexed and carboplatin
  2. Radiation
  3. Participants evaluated for response
  4. Lobectomy surgery
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Radiation: Radiation Therapy; Procedure: Lobectomy
- Arm B (Experimental): 1. Patients will be given the drugs pemetrexed and cisplatin
  2. Radiation
  3. Participants evaluated for response
  4. Lobectomy surgery
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Radiation: Radiation Therapy; Procedure: Lobectomy

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed by vein every 21 days for 3 cycles
  Arms: Arm A
Drug: Carboplatin — Carboplatin by vein Every 21 days for 3 cycles
  Arms: Arm A
Radiation: Radiation Therapy — Radiation treatment 5 days a week for 5-6 weeks.
  Arms: Arm A
Drug: Pemetrexed — Pemetrexed by vein every 21 days for 3 cycles
  Arms: Arm B
Drug: Cisplatin — Cisplatin by vein every 21 days for 3 cycles
  Arms: Arm B
Radiation: Radiation Therapy — Radiation treatment 5 days a week for 5-6 weeks.
  Arms: Arm B
Procedure: Lobectomy — Surgery
  Arms: Arm A
Procedure: Lobectomy — Surgery to remove a portion of the lung where the tumor is located.
  Arms: Arm B

SUMMARY:
This study is open to patients that have been diagnosed with non-squamous Stage III Non Small Cell Lung Cancer (NSCLC) and will have surgery to remove the tumor.

The purpose of this study is to:

* Test a combination of two chemotherapeutic drugs along with radiation therapy, when given prior to surgery and see what effects (good or bad) it has on someone with this type of cancer. Chemotherapeutic drugs selectively destroy diseased cancer cells and tissues.
* Test the safety of different dose levels of radiation when given with each combination of chemotherapy;
* Determine what side effects are associated with combining radiation with these two chemotherapy combinations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed non-squamous NSCLC.
* Resectable T3, and or N2 disease (T3N1, and resectable T1-3N2 multi-station non-bulky with no nodal station being more than 2 cm on preoperative workup, T4N0-1
* Resectable T3 includes patients with a satellite lesion in the same lobe as the primary.
* Male or Female, aged > or = 18 years and be able to give informed consent.
* Tumor should be technically operable with a lobectomy, bilobectomy or a sleeve resection.
* Patient should be medically operable
* ECOG Performance Status 0 or 1.
* Adequate bone marrow, hepatic and renal function assessed within 28 days
* Signed informed consent.
* Women of childbearing potential should have negative pregnancy test prior to enrollment to study.
* Men with partners in the childbearing age group and women of childbearing potential must use effective contraception while on treatment and for 6 months thereafter.
* The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed.
* The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.
* Patients must have a negative MRI or CT Scan of the brain.

Exclusion Criteria:

* Patients who have had chemotherapy or radiation therapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds or other agents used in study.
* Pregnant or lactating women.
* Male patients with female sexual partners in the reproductive age group who refuse to use effective methods of contraception will be excluded from the trial.
* Patients with concurrent serious infections.
* Patients with an unstable or serious concurrent medical condition are excluded.
* Presence of third space fluid which cannot be controlled by drainage.
* Weight loss > 10 percent from baseline weight.
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Patients with hypercalcemia will be excluded.
* Patients who require a pneumonectomy will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability
  Determine the safety and tolerability of concurrent chemotherapy with Cisplatin/ Pemetrexed or Carboplatin/Pemetrexed and dose escalated radiation therapy followed by lobectomy.

SECONDARY OUTCOMES:
Response rate, overall survival and progression free survival
  Evaluate the following:
  * Response Rate after concurrent chemoradiation therapy.
  * Overall Survival (OS).
  * Progression Free Survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States